CLINICAL TRIAL: NCT02099994
Title: A Phase I/IIa Clinical Trial of HIV-1 Vaccines pSG2.HIVconsv DNA, MVA.HIVconsv and Ad35-GRIN in Combined Regimens in Healthy HIV-1/2-negative Adults in Nairobi.
Brief Title: Safety & Immunogenicity of HIV Vaccines in Healthy Kenyan Adults
Acronym: HIV-CORE 004
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); International AIDS Vaccine Initiative (Network); Karolinska Institutet (Other); University of Nairobi (Other); Ichor Medical Systems Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIV-CORE 004/IAVI N004
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: AIDS
Keywords: HIV; vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - AM (Experimental): Ad35-GRIN 5 x 10^10 vp IM at week 0, MVA.HIVconsv 2 x 10^8 pfu IM at week 8.
  Interventions: Biological: Ad35-GRIN; Biological: MVA.HIVconsv
- B - DDDAM (Experimental): pSG2.HIVconsv DNA 4 mg or saline placebo at weeks 0, 4 and 8. Ad35-GRIN 5 x 10^10 vp or saline placebo at week 12. MVA.HIVconsv 2 x 10^8 pfu or saline placebo at week 20.
  Interventions: Biological: Ad35-GRIN; Biological: MVA.HIVconsv; Biological: pSG2.HIVconsv DNA
- C - DeDeDeAM (Experimental): Electroporated pSG2.HIVconsv 4 mg or electroporated saline placebo at weeks 0, 4 and 8.
  Ad35-GRIN 5 x 10^10 vp or saline placebo at week 12. MVA.HIVconsv 2 x 10^8 pfu or saline placebo at week 20.
  Interventions: Biological: Ad35-GRIN; Biological: MVA.HIVconsv; Biological: Electroporated pSG2.HIVconsv

INTERVENTIONS:
Biological: Ad35-GRIN — intramuscular administration of Ad35-GRIN 5 x 10^10 vp or saline placebo
Biological: MVA.HIVconsv — IM administration of MVA.HIVconsv 2 x 10^8 pfu or saline placebo
Biological: pSG2.HIVconsv DNA — IM administration of pSG2.HIVconsv DNA 4 mg or saline placebo
  Arms: B - DDDAM
Biological: Electroporated pSG2.HIVconsv — IM administration of electroporated pSG2.HIVconsv 4mg or saline placebo
  Arms: C - DeDeDeAM

SUMMARY:
The study is part of a long-term aim to develop an effective HIV-1 vaccine and will evaluate safety and immunogenicity of vaccines focusing T cell responses on the conserved region of the HIV-1 proteome. The vaccines used are pSG2.HIVconsv DNA (D), MVA.HIVconsv (M) and Ad35-GRIN (A), delivered in regimens AM, DDDAM and DeDeDeAM, where e indicates electroporation.

DETAILED DESCRIPTION:
The main objectives of this study are to determine the vaccines' safety and immunogenicity in an African population, and further strengthen the vaccine trial capacity in the South.

HIV-CORE 004 is a double blind, placebo controlled randomized Phase I/IIa study designed to evaluate the safety and immunogenicity of different delivery regimens using three novel HIV-1 vaccines pSG2.HIVconsv DNA (D) with and without electroporation (e), adenovirus Ad35-GRIN (A) and poxvirus MVA.HIVconsv (M) administered by intramuscular needle injection in heterologous prime-boost regimens.

72 healthy, low-risk, HIV-1-uninfected adult volunteers in Nairobi will be randomly assigned to one of three groups, AM, DDDAM and DeDeDeAM each containing 20 vaccinees and 4 placebo recipients.

Firstly, this study aims to evaluate the safety and tolerability of the vaccines pSG2.HIVconsv DNA (D) with and without electroporation (e), adenovirus Ad35-GRIN (A) and poxvirus MVA.HIVconsv (M).

Secondly, we shall determine the effect of electroporation during DNA priming on the frequency, durability and/or quality of T cell responses (DDDAM vs DeDeDeAM).

Thirdly, we shall determine whether priming with three DNA vaccinations with or without electroporation affects the frequency, durability and/or quality of T cell responses to the HIVconsv immunogen compared to that seen in the AM regimen (AM vs DDDAM/DeDeDeAM).

As this is the first study of the combined HIVconsv vaccines in an African population, of the pSG2.HIVconsv DNA with electroporation, and the combination of the two HIVconsv vaccines with Ad35-GRIN, this trial has been designed as a pilot study to compare different vector combinations. The sample sizes will only allow detection of large response differences between volunteers in the three groups, thus, yielding data that are primarily descriptive.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-50
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* Written informed consent.
* Willing to undergo HIV-1 testing, counselling and receive test results.
* All female volunteers must be willing to undergo urine pregnancy tests
* If sexually active using an effective method of contraception until at least 4 months after the last vaccination.
* Willing to forgo donating blood during the study.

Exclusion Criteria:

* Any relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease, or use of systemic corticosteroids, immunosuppressive, antiviral, anticancer or other medication that, in the opinion of the Principal Investigator or designee, is clinically significant, within the previous 6 months. (Note: use of inhaled steroids for asthma or use of topical steroids for localized skin conditions will not exclude a volunteer from participation.)
* Any clinically significant acute or chronic medical condition that is considered progressive or, in the opinion of the Principal Investigator or designee, would make the volunteer unsuitable for the study.
* Any of the following abnormal laboratory parameters (1 abnormal test may be repeated once if thought to be due to a temporary condition):

  * Haematology

    * Haemoglobin < 9.0 g/dl for women and <11.0 g/dl for men
    * Absolute Neutrophil Count (ANC) ≤ 1000 /mm3 (≤ 1 x 109 /l)
    * Absolute Lymphocyte Count (ALC) ≤ 600 /mm3 (≤0.6 x 109 /l)
    * Platelets ≤100,000 /mm3, ≥ 550,000 /mm3 (≤ 100 /l, ≥ 550 /l)
  * Biochemistry

    * Creatinine > 1.3 x upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) > 2.5 x ULN
    * Alanine aminotransferase (ALT) > 2.5 x ULN
  * Urinalysis- Clinically significant abnormal dipstick confirmed by microscopy:

    * Protein = 2+ or more
    * Blood = 2+ or more (for women: before or after menses)
* Confirmed HIV-1 or HIV-2 infection.
* If female, pregnant or planning a pregnancy any time from enrolment to 4 months after the last vaccination; or lactating.
* Receipt of live attenuated vaccine within the previous 60 days or planned receipt at any time until 60 days after vaccination with Investigational Medicinal Product (IMP) or receipt of other vaccine, including influenza vaccine, within the previous 14 days or planned receipt at any time until 14 days after vaccination with the IMP.
* Receipt of blood transfusion or blood products within the previous 6 months.
* Participation in another clinical trial of an IMP currently or within the previous 3 months or expected participation during this study.
* Receipt of any investigational HIV-1 vaccine within the last 6 years.
* History of severe or very severe local or systemic reactogenicity events after vaccination, or history of severe or very severe allergic reactions.
* Confirmed diagnosis of acute or chronic hepatitis B virus infection (spontaneous clearance leading to natural immunity, indicated by antibodies to core + antigens, is not an exclusion criterion); confirmed diagnosis of hepatitis C virus infection; untreated syphilis.
* Smallpox vaccination within the previous 3 years.
* Major psychiatric illness in the previous 3 years.
* History of allergy or hypersensitivity to latex, chronic skin problems such as eczema or psoriasis, or skin and subcutaneous tissue thickness > 40 mm as assessed by skin pinch test in either deltoid region.
* Presence of an implantable device
* Current use of any electronic stimulation device. Therapeutic or traumatic metal implant in either deltoid region.
* History of, or known active cardiac disease or a heart condition under the care of a doctor. Note: Slight physiological variation of normal resting heart rate (60 - 100 beats/minute) with respiration is NOT excluded.
* History of syncope or fainting episode within 1 year of study entry.
* Seizure disorder or any history of prior seizure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Vaccine Safety | 44 weeks
  Proportion of volunteers who develop a grade 3 or 4 local reaction. Proportion of volunteers who develop a grade 3 or 4 systemic reaction

SECONDARY OUTCOMES:
Vaccine immunogenicity | 44 weeks
  T cell responses will be determined initially by interferon-gamma enzyme-linked immunospot assay
Vaccine Safety | 44 weeks
  A descriptive summary of grade 3 of 4 local and systemic events including laboratory abnormalities.
  A descriptive summary of serious adverse events, including laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Walter Jaoko, Principal Investigator — University of Nairobi
Locations (1):
- KAVI-Kangemi clinic, Nairobi, Kenya